CLINICAL TRIAL: NCT07058454
Title: Development of an Active Surveillance System for Adverse Reactions to Molecular Targeted Drugs Based on Biomarkers and Personalized Medicine and Its Impact on Patient Quality of Life
Brief Title: Multicenter Prospective Observational Study of Cardiotoxicity in Patients Receiving Targeted Cancer Therapies
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024ZSLYEC-667
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-06

CONDITIONS: Cancer;Cardiovascular;Adverse Events; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood for genomic analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with Cardiovascular Adverse Events (MACE Group).: Participants who experience one or more major adverse cardiovascular events during the study period. This case group will consist of all patients in the cohort who develop a new cardiovascular event (e.g., heart failure, arrhythmia, myocardial ischemia, thromboembolism, etc.) while undergoing chemotherapy or by the end of follow-up.
- Group 2: Patients without Cardiovascular Adverse Events (No MACE Group).: Participants who do not experience any major cardiovascular adverse event during the study period. This control cohort includes patients from the same population (cancer patients on chemo/targeted therapy) who complete their treatment and follow-up without incident MACE. These patients will be frequency-matched by general characteristics such as age and sex to the MACE group for comparisons (all are adult Chinese patients with malignancy, no history of prior thrombotic events).

SUMMARY:
This study will prospectively monitor cancer patients receiving chemotherapy (including molecular targeted therapies) for cardiovascular adverse events using biomarkers and imaging. The goal is to develop a predictive model for major adverse cardiovascular events (MACE) in this population by integrating both local factors (e.g. central venous catheter-related thrombosis) and systemic factors (e.g. age, comorbidities, genetic predisposition). An active surveillance system employing periodic cardiac evaluations (ECG, echocardiography) and biomarker measurements (troponin T, NT-proBNP) will enable early detection of cardiotoxic effects. The impact of these adverse events and the monitoring strategy on patients' quality of life will also be assessed.

DETAILED DESCRIPTION:
Cancer patients are at heightened risk of cardiovascular complications due to both their disease and its treatments. Many chemotherapeutic and targeted agents (e.g. anthracyclines, trastuzumab, bevacizumab, tyrosine kinase inhibitors) carry cardiotoxic potential, leading to diverse manifestations of MACE such as heart failure, arrhythmias, ischemic heart disease, valvular dysfunction, hypertension, thromboembolism, and others. As cancer survival improves and newer therapies are widely used, the incidence of treatment-related cardiac toxicity continues to rise. Early cardiotoxic changes are often subclinical, making proactive monitoring essential. Research has shown that cardiac biomarkers can rise before left ventricular ejection fraction declines, enabling "pre-symptomatic" detection of cardiotoxicity. By quantitatively analyzing the predictive value of each indicator for MACE, the study aims to construct a comprehensive risk prediction model for precise cardiovascular risk evaluation in cancer patients. Both local risk factors (e.g., indwelling catheter-related thrombosis) and systemic factors (e.g., age, hypercoagulability, body mass index) will be incorporated, reflecting the interplay of factors contributing to MACE. Genetic biomarkers will also be explored: blood samples are collected for genomic analysis (such as SNP genotyping and whole genome sequencing) to identify genetic polymorphisms associated with increased susceptibility to therapy-related MACE. By comparing patients who develop cardiovascular events to those who do not, we will characterize the incidence, timing, affected organs, and clinical presentation of MACE in cancer patients. Patient-reported quality of life will be evaluated using validated questionnaires, to determine how the occurrence of adverse cardiovascular events (and the implementation of active monitoring) affects daily functioning and overall well-being. Ultimately, this study's findings will provide a scientific basis for individualized risk stratification and preventive interventions in cardio-oncology, supporting optimized clinical strategies to mitigate cardiovascular risk without compromising effective cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1.Adults (age > 18 years) with a pathologically confirmed malignant tumor (any type of cancer); 2.Currently receiving or planning to receive chemotherapy (including regimens containing molecular targeted drugs) as adjuvant treatment for cancer; 3.Willing and able to participate in the study with provision of informed consent, and agreeable to provide required clinical data and biological samples.

-

Exclusion Criteria:

1. Incomplete basic patient information or medical records (missing key data necessary for the study);
2. Failure to complete the full course of planned chemotherapy at the study center (e.g., patient did not adhere to or finish all cycles of adjuvant chemotherapy at our institution);
3. History of severe acute cardiovascular or cerebrovascular events within 6 months prior to enrollment, including acute heart failure, acute myocardial infarction, acute intracerebral hemorrhage (stroke), malignant arrhythmia, or New York Heart Association (NYHA) Class IV/V heart failure;
4. Missing essential pre- or post-chemotherapy evaluations: patients who did not undergo complete baseline or end-of-treatment assessments (such as blood routine, hepatic/renal function, coagulation profile, cardiac enzymes (troponin T), NT-proBNP (or BNP), 12-lead ECG, and echocardiogram)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult cancer patients receiving adjuvant chemotherapy (including those receiving molecular targeted agents as part of therapy) at included centers (and collaborating centers) between June 1, 2025 and June 30, 2027. Eligible patients include those with any malignant solid tumor or hematologic malignancy who are starting a planned course of postoperative (adjuvant) chemotherapy. Enrollment will be consecutive and non-selective - all patients meeting inclusion criteria (and no exclusion criteria) in the participating centers during the accrual window will be invited to participate. Patients are typically enrolled at the time of initiation of chemotherapy, with baseline cardiovascular assessments performed prior to or at the first cycle of treatment. The cohort will be followed prospectively through their chemotherapy course and for up to 6 months after completion of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of New Onset Major Adverse Cardiovascular Events (MACE) by End of Chemotherapy | From initiation of chemotherapy to end of adjuvant chemotherapy (approximately up to 6 months per patient).
  Occurrence of any new cardiovascular adverse event from start of chemotherapy to the completion of the chemotherapy regimen. "MACE" is defined per ESC guidelines to include major cardiac events such as new myocardial dysfunction, symptomatic heart failure, coronary artery disease (e.g. myocardial infarction), clinically significant valvular disease, arrhythmia (e.g. atrial fibrillation), new or worsening hypertension, thromboembolic events (including deep vein thrombosis or pulmonary embolism), peripheral vascular disease, pulmonary hypertension, or pericardial disease. Any such event recorded on electrocardiogram, cardiac ultrasound (echocardiography), or via cardiac enzymes (troponin T) and biomarkers (NT-proBNP/BNP) by the end of the adjuvant chemotherapy cycle, relative to the patient's pre-treatment baseline, will be counted as an outcome event. (Early cardiovascular events are defined as those occurring during the chemotherapy period.)

SECONDARY OUTCOMES:
Quality of Life Score Change (Baseline to 6 Months Post-treatment) | Baseline pre-therapy and 6 months after completion of chemotherapy.
  Change in patient-reported quality of life from baseline (pre-therapy) to follow-up after therapy completion. Quality of life will be measured using a validated questionnaire (e.g., EORTC QLQ-C30 or similar cancer-specific QoL instrument) at study entry and at 6 months after the last chemotherapy cycle. The difference in global health/QoL scores and functional subscales will be analyzed to determine the impact of any adverse events and the monitoring program on patients' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: xiaoyan li, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No